CLINICAL TRIAL: NCT00580580
Title: The Detection of Coronary Stenosis With Intravenous Mircrobubbles and Contrast Pulse Sequence Low Mechanical Index Imaging
Brief Title: Detection of Coronary Stenosis With Intravenous Microbubbles
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0060-03-FB
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Coronary Stenosis; Carotid Stenosis; Myocardial Reperfusion
MeSH Terms: conditions — Coronary Stenosis; Carotid Stenosis | interventions — FS 069; perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 Intravenous Optison Followed by Contrast Pulse Sequencing (Active Comparator): Administration of Optison (0.1-0.4 mL) intravenously followed by Contrast Pulse Sequencing to image both the coronary and carotid arteries.
  Use will depend on availability of the contrast for the given study Optison will not be used on patients with blood allergies or Jehovah Witnesses
  Interventions: Drug: Optison
- 2 Intravenous Definity followed by Contrast Pulse Sequencing (Active Comparator): Intravenous injection of Definity (0.05-0.20 mL) followed by Contrast Pulse Sequencing to image both coronary and carotid arteries
  Interventions: Drug: Definity
- 3 Intravenous PESDA followed by Contrast Pulse Sequencing (Active Comparator): Intravenous injection of PESDA at a rate of 0.05-0.20 mL followed by Contrast Pulse Sequencing image of coronary and carotid arteries PESDA will be used exclusively in patients who are eligible for other IRB studies
  Interventions: Drug: PESDA

INTERVENTIONS:
Drug: Optison — 0.1-0.4 mL through intravenous injection at the beginning of the study.
  Arms: 1 Intravenous Optison Followed by Contrast Pulse Sequencing
Drug: Definity — intravenous injection at 0.05-0.20 mL
  Arms: 2 Intravenous Definity followed by Contrast Pulse Sequencing
Drug: PESDA — intravenous injections dosage 0.05-0.20 mL
  Other Names: PESDA is an investigational drug (IND 54,263)
  Arms: 3 Intravenous PESDA followed by Contrast Pulse Sequencing

SUMMARY:
To detect coronary artery disease by both coronary and carotid artery imaging and myocardial perfusion imaging using a new low mechanical index real time system.

DETAILED DESCRIPTION:
The objective of this clinical study will be to visualize both coronary and carotid arteries as well as detect myocardial perfusion following a routine intravenous injection of Definity (0.05-0.20 millimeters), Optison (0.1-0.4 millimeters) or PESDA (0.05-0.2 mL). Following these injections , we will attempt to Contrast Pulse Sequencing on the Siemens Acuson Sequoia system to image both the coronary and carotid arteries, as well as the Myocardial perfusion.

ELIGIBILITY:
Inclusion Criteria:

* subjects scheduled for routine echocardiogram to look for evidence of Coronary artery disease or a stress echocardiogram
* women of child-bearing potential must be taking a medically approved form of birth control with a negative urine pregnancy test
* be conscious and coherent, and be able to communicate effectively with study personnel
* last eight patients will be diabetics who smoke
* provide informed consent after receiving a verbal and written explanation of the purpose and nature of the study

Exclusion Criteria:

* severe valvular heart disease by Doppler Echocardiography
* females of child-bearing potential who are not taking a medically approved method of birth control will be excluded. If the patient is pregnant she will be excluded.
* patients who are allergic to blood or blood products will be excluded
* have contraindication to Optison, Definity, or PESDA (pulmonary HTN, cardiac shunt)
* non diabetics, non smokers

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Detection of coronary and carotid artery stenoses and perfusion defects during standard echocardiographic examination | 2-4 months
  To determine whether this imaging scheme can detect both coronary and carotid artery stenoses as well as perfusion defects during a standard echocardiographic examination

SECONDARY OUTCOMES:
Visual analysis of coronary and carotid arteries and perfusion defects during standard echocardiogram examination | immediate
  Visually analyze the coronary and carotid arteries as well as perfusion defects during a standard echocardiogram examination

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Porter, MD, Principal Investigator — University of Nebraska